CLINICAL TRIAL: NCT00991978
Title: Vascular Endothelial Growth Factor (VEGF) Imaging for Early Breast Cancer Detection A Feasibility Study
Brief Title: VEGF Early Imaging for Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, C.P. Schroder, dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VEGF early imaging
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; VEGF; Screening
MeSH Terms: conditions — Breast Neoplasms | interventions — 89Zr-bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 89Zr-bevacizumab PET (Experimental): 89Zr-bevacizumab PET
  Interventions: Other: 89Zr-bevacizumab PET

INTERVENTIONS:
Other: 89Zr-bevacizumab PET — PET-scan with 89Zr-bevacizumab
  Other Names: 89Zr-bevacizumab

SUMMARY:
Breast cancer is the most common cause of cancer death among women. Yearly around 12,500 Dutch women are diagnosed with breast cancer and 3,500 die of this disease. One of the problems leading to such striking effect refers to late tumor detection due to inadequate sensitivity of current imaging techniques. Current screening is performed by means of mammography, consisting of traditional film-screen mammograms of digital mammograms. These digital mammograms offer digital enhancement to aid interpretation, which is especially helpful in women with dense breast tissue. Screening mammography is nowadays the single most effective method of early breast cancer detection. For screening of high risk individuals, increasingly the magnetic resonance imaging (MRI) technique is emerging. However, none of the above mentioned techniques has an optimal sensitivity and specificity, leading for instance to a significant portion of false positive results. The clinical consequence of this error is that additional tests and procedures are performed in women who may not have cancer. In the United States, for example, 11% mammograms require additional evaluation; the lesion turns out to be benign in more than 90% of cases [1].

False-positive readings False positive readings are more common in younger women, both because the tests are less specific and because breast cancer is less common [2,3]. As a result, more follow-up procedures, including invasive procedures such as biopsies, will be done in younger women even though fewer cancers will be found. Furthermore, because breast cancer screening occurs repeatedly, the risk of a false-positive study is likely to rise with repeated screening [4].

Emerging adjuncts to mammography include ultrasonography, which is helpful for further assessment of known areas of interest, and magnetic resonance imaging. Image-guided biopsy - directed by ultrasonography or stereotactic mammography views - plays a critical role in histological confirmation of suspected breast cancer.

DETAILED DESCRIPTION:
Objectives of the trial

Primary objective The aim is to perform a feasibility study to show that VEGF PET imaging using 89Zr-bevacizumab as tracer can be used for early breast cancer detection.

Secondary Objectives A secondary aim is whether positive lymph nodes can be detected.

End-points

* The primary endpoint will be 89Zr-bevacizumab tracer uptake in primary breast tumors < 2 cm.
* The secondary endpoint will be 89Zr-bevacizumab tracer uptake in axillary lymph nodes.

Patient selection criteria

Inclusion

* Patients with a breast tumor size < 2 cm in diameter (as determined by means of conventional imaging techniques: mammography, ultrasound or MRI) who are scheduled to receive operative intervention either by means of a mastectomy or lumpectomy.
* histologically proven breast cancer
* Age > 18 years.
* WHO performance status 0-2 (see: appendix B)
* Signed written informed consent (approved by the Institutional Review Board [IRB]/ Independent Ethics Committee [IEC]) obtained prior to any study specific screening procedures.
* Able to comply with the protocol.

Exclusion

* Other invasive malignancy or condition which could affect compliance with the protocol or interpretation of results.
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for pre-menopausal women with intact reproductive organs and for women less than two years after menopause.
* Prior radiotherapy on the involved area.
* Major surgery within 28 days before the initiation of the study.
* Clinically significant cardiovascular disease.
* Prior allergic reaction to immunoglobulins or immunoglobulin allergy.

Trial Design All patients will undergo a 89Zr-bevacizumab PET scan preoperatively at day 4 following tracer injection (see: section 16 for timetable). The uptake of 89Zr-bevacizumab in the tumor will be quantified. Results will be fused and compared with standard imaging techniques and with standard tumor histology as well as specific tumor stainings for angiogenesis including VEGF staining. Sensitivity and specificity will be compared with conventional imaging.

Study assessments

89Zr-bevacizumab PET imaging

Radiolabelling of bevacizumab Conjugation and radiolabeling of the monoclonal antibody is essentially performed as has been described by Verel et al (15), with only minor adjustments with regard to purification. In short: FTP-N-sucDf-Fe (kindly provided by the VU University Medical Center, Amsterdam, The Netherlands) was conjugated to the mAb at a 10:1 molar ratio. Fe(III) is subsequently removed by an excess of EDTA (Calbiochem, San Diego, California, USA) for 30 min at 35°C and the antibody is purified by ultrafiltration (Vivaspin-2 Centrifugal Concentrator, filter 30 kDa, Sartorius, Göttingen, Germany). This purified antibody is either stored at -80°C or immediately used for radiolabelling. The conjugated antibody is added to 89Zr-oxalate (100-1000 MBq/mg mAb, kindly provided by the VU University Medical Center, Amsterdam, The Netherlands), 0.9% NaCl (Braun Melsungen AG, Oss, The Netherlands), 2M Na2CO3 (OPG Farma, Utrecht, The Netherlands) and 0.5M HEPES buffer (Sigma-Aldrich, Zwijndrecht, The Netherlands). After 60 minutes, the radiolabeled antibody is purified by ultrafiltration Vivaspin-2 Centrifugal Concentrator, filter 30 kDa, Sartorius, Göttingen, Germany) and diluted in 0.9% NaCl/gentisic acid (5 mg/ml, Merck Schuchardt OHG, Hohenbrunn, Germany). The 89Zr isotope has a physical t ½ of 78 hours. 89Zr-bevacizumab has radiochemical purity >95% and excellent long term stability in human serum (> 1 week). Conjugation and radiolabeling is performed in the radiopharmacy facilities of the department of Nuclear Medicine and Molecular Imaging under GMP-conditions, under responsibility of a hospital pharmacist. More detailed information regarding 89Zr-bevacizumab is found in the investigational medicinal medicinal product dossier (IMPD; appendix C).

PET imaging Patients will be injected intravenously with 37 MBq 89Zr-bevacizumab (protein dose 5 mg) at day 0. Subsequently, images will be made 4 days after the injection of 89Zr-bevacizumab (see section 16 for timetable). For imaging a Siemens PET/CT camera will be used. Recording will be performed in 3D mode from lower thorax to neck, in approximately 2 bedpositions. The Department of Nuclear Medicine and Molecular Imaging is certified according to the ISO-NEN-9001 standard. Standard operating procedures for dynamic scanning will be used for all PET scans. Actual operation of the PET camera and scan acquisition will be performed by a nuclear medicine technologist. Final image analysis will be performed by a nuclear medicine specialist. 89Zr-bevacizumab distribution will be scored visually and quantitatively.

The majority of patients will also undergo sentinel node detection for staging of the axilla during the surgical treatment of the primary tumor. For the sentinel node procedure, 99mTechnetium labeled nanocolloid is used. The anticipated time between 89Zr-bevacizumab and 99mTc-nanocolloid administration will be approximately 2 weeks. By then, 7 half-life episodes of the 89Zr radiolabel will have passed and its signal will be negligible. Therefore, no interference of the radiolabel signals is expected.

Radiation dose/safety Use of positron emitting isotopes means exposure to ionizing radiation. Because of the potential hazards of radiation, guidelines for the exposure of healthy volunteers are specified in "Besluit Stralingsbescherming (BS 2000), artikel 64 - en Nota van Toelichting (Staatsblad 2001, 397)", which refers to the guidelines of the International Commission on Radiological Protection (ICRP). As the kinetics of the antibody bevacizumab are almost comparable to those of trastuzumab, the radiation dose of 89Zr labelled bevacizumab is expected to be in the same range as that of 89Zr-trastuzumab.

For estimating the radiation dose to a 'standard female' during 89Zr-trastuzumab scanning, use was made of available kinetic data from previous 111In-trastuzumab planar imaging. This is possible as the halftime of 111In is in the same order of magnitude as that of 89Zr and therefore it enables us to track tracer kinetics over a time period that is also relevant for 89Zr dosimetry. Using scan-series consisting of 4 consecutive planar scans over a period of 168 hours, residence times of the main source organs and the whole-body were calculated, adjusting for the difference in nuclide half-lives. These residence times were fed into the OLINDA program, which calculates the effective radiation dose using the MIRD scheme. The final estimate was found from averaging the results from 5 different patients, yielding 18 mSv for an injected dose of 37 MBq. In the current protocol, this would result in a radiation dose (including the attenuation correction for low dose CT) of 19.5 mSv for women (and 16.5 mSv for men). According to ICRP 62 this radiation dose falls in category III (moderate risk).

Tumor staining In addition to the standard evaluation of the postoperative tumor specimen, specific staining for VEGF pathway related proteins will be performed including VEGF, CD34 staining for mean vascular density (MVD), SMA for vascular maturation, HIF-1alpha for hypoxia, VEGF receptors, Ki 67 for proliferation or other relevant staining according to the most up to date scientific insights.

Clinical evaluation, laboratory tests, follow- up

Before start

* Physical examination
* WHO performance score (see appendix B)
* Conventional imaging of the breast (mammography, ultrasound or MRI)
* Histological confirmation of malignant breast lesion
* Evaluation of in- and exclusion criteria
* Signed written informed consent

Criteria of evaluation

PET scan PET scans will be evaluated by a nuclear medicine physician blinded for clinical information and location of the tumor. The PET data will be correlated to the conventional imaging data. The final postoperative pathological evaluation will be related to the PET data.

Tumor staining Evaluation of VEGF related tumor staining will be performed in collaboration with a pathologist, blinded for clinical information.

Statistical considerations

In this feasibility study we will postulate high demands to prove the sensitivity of 89Zr-bevacizumab-PET scan to detect breast cancer lesions in order to justify our final future aim to obtain a good discrimination between benign versus pre-malignant/malignant lesions with VEGF imaging. Demands for very high sensitivity to detect the tumor with 89Zr-bevacizumab-PET scanning requires a sensitivity no worse than 99%.

We will use a stopping rule with a type 1 error of 5% (one-sided alpha of 5%) and a beta of 10% (~a power of 90%), and external reference values for false negative rates of 0.01 and as alternative 0.10. An extensive description of the stopping rule with two boundaries, is included in appendix C.

In the present study, the requirements are p0=0.01, p1=0.10, alpha(rule)=0.05, beta(rule)=0.10 and alpha(futile)=0.05. After exact calculation, this results in alpha(n)=0.1364, beta(N)=0.055 and alpha(futile,n)=0.6431, with 47 as the maximum number of patients. With a true failure rate of 0.01, the probability of passing the upper boundary is 0.049; with a true failure rate of 0.10 this probability is 0.903. The upper boundary, representing the maximum of acceptable failures, is 1 within the first 35 patients and 2 up to the total number of 47 patients. Monitoring with the stopping rule can be stopped (because of futile testing) when no failures are observed within the first 31 patients.

Investigator authorization procedure

The specialist who will treat the patient or his/her research nurse can sign up a patient for registration.

Patient registration

To enter patients in this study, during working hours, the data manager should be contacted at:

University Medical Centre Groningen Department of Medical Oncology Phone: 050-3612053 or page nr 77045 Eligibility will be checked at the time of registration.

To determine eligibility the following information should be provided:

* Initials
* Date of birth
* WHO performance score
* Signed written informed consent
* Date of intended surgery (if known)

Forms and procedures for collecting data

Data will be collected on paper case record forms (CRF). CRFs will be collected and data will be entered anonymously in an Access data base.

Subject identification Patient data are stored under a code without name, that will ensure anonimity.

Informed consent All patients will be informed of the aims of the study, the possible adverse events, the procedures and possible hazards to which he/she will be exposed, and the mechanism of treatment allocation. They will be informed as to the strict confidentiality of their patient data, but that their medical records may be reviewed for trial purposes by authorized individuals other than their treating physician. An example of a patient informed consent statement is given as an appendix to this protocol.

The ethics committee of the UMCG will validate local informed consent documents before start of the study.

It will be emphasized that the participation is voluntary and that the patient is allowed to refuse further participation in the protocol whenever he/she wants. This will not prejudice the patient's subsequent care. Documented informed consent must be obtained for all patients included in the study before they are registered or randomized in the study. This must be done in accordance with the national and local regulatory requirements.

The informed consent procedure must conform to the ICH guidelines on Good Clinical Practice. This implies that "the written informed consent form should be signed and personally dated by the patient or by the patient's legally acceptable representative".

ELIGIBILITY:
Inclusion Criteria:

* Patients with a breast tumor size < 2 cm in diameter (as determined by means of conventional imaging techniques: mammography, ultrasound or MRI) who are scheduled to receive operative intervention either by means of a mastectomy or lumpectomy.
* histologically proven breast cancer
* Age > 18 years.
* WHO performance status 0-2 (see: appendix B)
* Signed written informed consent (approved by the Institutional Review Board [IRB]/ Independent Ethics Committee [IEC]) obtained prior to any study specific screening procedures.
* Able to comply with the protocol.

Exclusion Criteria:

* Other invasive malignancy or condition which could affect compliance with the protocol or interpretation of results.
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for pre-menopausal women with intact reproductive organs and for women less than two years after menopause.
* Prior radiotherapy on the involved area.
* Major surgery within 28 days before the initiation of the study.
* Clinically significant cardiovascular disease.
* Prior allergic reaction to immunoglobulins or immunoglobulin allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
SUV in tumour and lymph nodes | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Schröder, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Universitar Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Brown ML, Houn F, Sickles EA, Kessler LG. Screening mammography in community practice: positive predictive value of abnormal findings and yield of follow-up diagnostic procedures. AJR Am J Roentgenol. 1995 Dec;165(6):1373-7. doi: 10.2214/ajr.165.6.7484568.
- [Background] Kerlikowske K, Grady D, Barclay J, Sickles EA, Eaton A, Ernster V. Positive predictive value of screening mammography by age and family history of breast cancer. JAMA. 1993 Nov 24;270(20):2444-50. PMID 8230621
- [Background] Lidbrink E, Elfving J, Frisell J, Jonsson E. Neglected aspects of false positive findings of mammography in breast cancer screening: analysis of false positive cases from the Stockholm trial. BMJ. 1996 Feb 3;312(7026):273-6. doi: 10.1136/bmj.312.7026.273. PMID 8611781
- [Background] Eddy DM. Screening for breast cancer. Ann Intern Med. 1989 Sep 1;111(5):389-99. doi: 10.7326/0003-4819-111-5-389. PMID 2504094
- [Background] Sledge GW Jr. VEGF-targeting therapy for breast cancer. J Mammary Gland Biol Neoplasia. 2005 Oct;10(4):319-23. doi: 10.1007/s10911-006-9005-5. PMID 16924373
- [Background] Kataoka N, Cai Q, Wen W, Shu XO, Jin F, Gao YT, Zheng W. Population-based case-control study of VEGF gene polymorphisms and breast cancer risk among Chinese women. Cancer Epidemiol Biomarkers Prev. 2006 Jun;15(6):1148-52. doi: 10.1158/1055-9965.EPI-05-0871. PMID 16775174